CLINICAL TRIAL: NCT01409447
Title: Repair of Articular Osteochondral Defect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ching-Chuan Jiang, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200707007D
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Osteochondritis Dissecans
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biphasic osteochondral composite (Experimental): feasibility study for the new medical device & technique
  Interventions: Device: Biphasic osteochondral composite

INTERVENTIONS:
Device: Biphasic osteochondral composite — We had previously developed a biphasic osteochondral composite as the construct for chondrocyte implantation. We further conducted this feasibility study of such device to treat patients with osteochondral lesion of the knee joints.
  Other Names: Biphasic scaffold

SUMMARY:
Background: Matrix-associated autologous chondrocyte implantation (MACI) has been recently used to treat cartilage defects. The investigators had previously developed a biphasic osteochondral composite as the construct for chondrocyte implantation. The investigators further conducted this feasibility study of such device to treat patients with osteochondral lesion of the knee joints.

DETAILED DESCRIPTION:
Methods: Ten patients with symptomatic isolated osteochondritis at the femoral condyle were treated by replacing the pathological tissue with autologous chondrocyte-laden biphasic cylindrical plug of DL-poly-lactide-co-glycolide, with its lower body impregnated with -tricalcium phosphate as the osseous phase. The osteochondral lesion was drilled to fashion a pit of identical size and shape as the plug. The chondrocyte-laden plug was press-fit to fill the pit. Outcome of repair was examined by KOOS scale at 3, 6 and 12 months postoperatively, and tissue sample was collected with second-look arthroscopic needle-biopsy at 12 months. The primary outcome parameter was the postoperative change of KOOS; and the secondary outcome parameter was the regeneration of cancellous bone and hyaline cartilage at the repair site.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 ~ 60 years
* Articular cartilage defect of the knee
* Diagnosis by X-ray and/or MRI, Arthroscopy
* Confined area: diameter < 3 cm
* Full layer cartilage damage

Exclusion Criteria:

* Pregnancy
* Nonunion of fracture around the knee
* Diffuse degenerative arthropathy of the knee
* Diffuse cartilage pathology due to
* Rheumatism: rheumatoid, psoriatic, …
* Metabolic disorder: gouty, hemorrhagic, …
* Stiff knee from any reason
* Flexion < 130˚
* Extension loss > 20˚

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chuan Jiang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan